CLINICAL TRIAL: NCT04353921
Title: A Two-Year Observational Follow-up Study of Subjects With Major Depressive Disorder Following a Randomized, Double-Blind Single-Dose of Psilocybin or Niacin-Control
Brief Title: PSIL201 Long-term Follow-up Study: Psilocybin or Niacin / Major Depressive Disorder
Status: Terminated | Type: Observational
Why Stopped: Low enrollment and inability to achieve statistical significance
Sponsor: Usona Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PSIL201-LTFU
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single-Dose of Psilocybin
  Interventions: Other: No intervention will be administered as part of this study.
- Niacin-Control
  Interventions: Other: No intervention will be administered as part of this study.

INTERVENTIONS:
Other: No intervention will be administered as part of this study. — No intervention will be administered as part of this study.

SUMMARY:
This is a Phase 2 double-blind, long-term observational follow-up study of participants from Study PSIL201. Participants providing informed consent will be enrolled into this study and will complete web surveys and telephone interviews conducted by one central site at the following time intervals: months 2, 3, 4, 5 and 6 (± 7 days for each assessment) and months 8, 10, 12, 14, 16, 18, 20, 22 and 24 (± 14 days for each assessment).

ELIGIBILITY:
Inclusion Criteria:

* Enrollment and intervention with the investigational drug in Study PSIL201

Exclusion Criteria:

* Inability or unwillingness to complete study procedures, including regular completion of web surveys and telephone interviews with study personnel

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Enrollment is constrained to those participants dosed with investigational drug (psilocybin or niacin) in Study PSIL201.
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale | 6 Months post-dosing in PSIL201
  Between-group difference in mean change from baseline (prior to dosing in PSIL201) in Montgomery-Asberg Depression Rating Scale (MADRS)

CONTACTS AND LOCATIONS:
Locations (1):
- Segal Trials, Lauderhill, Florida, United States